CLINICAL TRIAL: NCT04376736
Title: SNAP HOME: Smart No-show Analytics Paired With Home-based Outpatient Medical Engagement
Brief Title: Home Visits for Patients at Risk for Appointment No-shows
Acronym: SNAP HOME
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical difficulties
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00196142
Record Dates: First submitted 2020-05-01; First posted 2020-05-06 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Utilization, Health Care; Engagement, Patient; No-Show Patients
MeSH Terms: conditions — Patient Acceptance of Health Care; Patient Participation; No-Show Patients | interventions — House Calls

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Patients are reminded about their appointments
- Intervention arm (Experimental): Patients are offered a one-time home visit by providers in lieu of their upcoming in-person visit
  Interventions: Other: Home visit

INTERVENTIONS:
Other: Home visit — Home visit by medical provider
  Arms: Intervention arm

SUMMARY:
Unused clinic visits due to patient no-shows continue to plague American healthcare as a large source of waste and avoidable constraint on access. The average no-show rate across 105 studies was 23% though with wide variation (4% to 79%). No-show behavior has adverse effects on patients, providers, and healthcare organizations' operational and financial outcomes. Patients that miss clinic visits are more likely to need acute care and suffer poor health outcomes. There have been increasingly sophisticated efforts focused on predicting which patients are likely to no-show. This can allow for tactful over-booking and/or patient outreach. At Hopkins, investigators have implemented a novel machine learning based approach for identifying those patients at high-risk for no-show. Offering home visits for patients who are most likely to no-show is an appealing strategy to connect medical providers with patients who need care but are otherwise unlikely to receive it. Yet, it is unclear if this would be helpful to engage patients in their care, and encourage subsequent attendance, or if it would encourage future missed appointments, fostering a reliance on possible ongoing home visits. This study would link existing efforts with no-show prediction to home visits by internal medicine residents and evaluate its clinical impact. Patients at high-risk for no-show will be randomized into the control arm where patients will be called to remind patients of their visits. Those randomized into the intervention arm will be offered a one time home visit in lieu of their in-person visit to help understand barriers to in-person care and build rapport. Outcomes evaluated include future in-person show rates and healthcare cost/utilization

ELIGIBILITY:
Inclusion Criteria:

* One or more poorly controlled chronic medical illness
* More than one chronic illness, regardless of its level of control
* Acute illness

Exclusion Criteria:

* No documented medical illnesses (acute or chronic)
* Single well controlled chronic illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Engagement | 1 year post enrollment
  Subsequent show up rate for medical clinic appointments, that is, number of actual visits per total number of expected visits

SECONDARY OUTCOMES:
Healthcare utilization as assessed by number of hospitalizations | 1 year post enrollment
  This will be assessed based on the Number of ER visits and hospitalizations

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No